CLINICAL TRIAL: NCT00756509
Title: An Open-label, Multi-center, Single-arm Study to Evaluate the Efficacy of Nilotinib in Adult Patients With Metastatic or Unresectable Gastrointestinal Stromal Tumors in First Line Treatment
Brief Title: Treatment of Patients With Metastatic or Unresectable Gastrointestinal Stromal Tumors in First Line With Nilotinib
Status: Completed | Phase: Phase 4 | Type: Interventional
Sponsor: Novartis Pharmaceuticals (Industry)
Responsible Party: Sponsor
Organization: Novartis (Industry)
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: CAMN107DDE06; 2008-000358-11 (EudraCT Number)
Record Dates: First submitted 2008-09-19; First posted 2008-09-22 (Estimated); Results first posted 2026-01-20 (Actual); Last update posted 2026-01-20 (Actual); Status verified 2026-01

CONDITIONS: Gastrointestinal Stromal Tumors
Keywords: unresectable or metastatic GIST; 1st. line treatment
MeSH Terms: conditions — Gastrointestinal Stromal Tumors | interventions — nilotinib

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- nilotinib (Experimental): nilotinib
  Interventions: Drug: Nilotinib

INTERVENTIONS:
Drug: Nilotinib — 800 mg/d orally

SUMMARY:
The purpose of this multicenter, single-arm, phase II trial is to evaluate the efficacy of Nilotinib in patients with unresectable or metastatic gastrointestinal stromal tumors (GIST).

DETAILED DESCRIPTION:
The study planned a 6-month recruitment phase to enroll 40 subjects, followed by a 6-month treatment phase with monthly visits. Patients benefiting from the treatment could continue during a follow-up phase.

On May 5, 2011, Novartis decided to discontinue the ongoing clinical trials with Nilotinib in GIST. This decision was influenced by the discontinuation of the ENESTg1 study (CAMN107G2301), which showed that Nilotinib was unlikely to demonstrate superiority to Imatinib in progression-free survival, the primary endpoint. The independent Data Management Committee (DMC) also reported no safety issues in either trial arm. Following the decision to close-out the Novartis- Sponsored studies CAMN107G2301 (NCT00785785) and CAMN107DDE05 (NCT01289028), the enrollment of the study CAMN107DDE06 was re-opened in order to ensure continued access to nilotinib to the patients currently in the CAMN107G2301 trial and CAMN107DDE05 trial in Germany and benefiting from the nilotinib treatment.

ELIGIBILITY:
Inclusion criteria

* Age ≥18 years
* Histologically confirmed diagnosis of GIST that is unresectable and/or metastatic and therefore not amenable to surgery or combined modality with curative intent prior to or at Visit 1
* At least one measurable site of disease on CT/MRI scan at Visit 1, as defined by RECIST criteria. The scans should be at maximum 2 weeks old. New scans are only required as baseline scans if they are older than approx. 2 weeks.
* WHO Performance Status of 0, 1 or 2
* Patients must have the following laboratory values (≥ LLN (lower limit of normal) or corrected to within normal limits with supplements prior to the first dose of study medication.):

  1. Potassium ≥ LLN,
  2. Magnesium ≥ LLN,
  3. Phosphorus ≥ LLN,
  4. Total calcium (corrected for serum albumin) ≥ LLN
* Patients must have normal organ, electrolyte, and marrow function as defined below:

  1. Absolute Neutrophil Count (ANC) ≥ 1.5x 109/L;
  2. Platelets ≥ 100 x 109/L;
  3. ALT and AST ≤ 2.5 x upper limit of normal (ULN) or ≤ 5.0 x ULN if considered due to tumor;
  4. Alkaline phosphatase ≤ 2.5 x ULN unless considered due to tumor;
  5. Serum bilirubin ≤ 1.5 x ULN;
  6. Serum lipase and amylase ≤ 1.5 x ULN;
  7. Serum creatinine ≤ 1.5 x ULN or 24-hour creatinine clearance ≥ 50 ml/min. (calculated creatinine clearance using Cockroft formula is acceptable)
* Ability to understand and willingness to sign a written informed consent

Exclusion criteria

* Prior treatment with nilotinib
* Treatment with any cytotoxic and/or investigational cytotoxic drug ≤ 4 weeks (6 weeks for nitrosurea or mitomycin C) prior to Visit 1 with the exception of imatinib targeted therapy as an adjuvant therapy or imatinib in first line treatment for maximum of 4 weeks.
* Prior or concomitant malignancies requiring active treatment other than GIST with the exception of previous or concomitant basal cell skin cancer, previous cervical carcinoma in situ
* Impaired cardiac function at including any one of the following:

  1. LVEF < 45% or below the institutional LLN range (whichever is higher) as determined by echocardiogram at Visit 1
  2. Complete left bundle branch block
  3. Use of a ventricular paced cardiac pacemaker
  4. Congenital long QT syndrome or family history of long QT syndrome
  5. History of or presence of significant ventricular or atrial tachyarrhythmias
  6. Clinically significant resting bradycardia (< 50 beats per minute)
  7. QTc > 450 msec on screening ECG (using the QTcF formula). If QTc > 450 msec and electrolytes are not within normal ranges (electrolytes should be corrected and then the patient rescreened for QTc.
  8. Right bundle branch block plus left anterior hemiblock, bifascicular block
  9. Myocardial infarction within 12 months prior to Visit 1
  10. Other clinically significant heart disease (e.g., unstable angina, congestive heart failure or uncontrolled hypertension,)
* Patients with severe and/or uncontrolled concurrent medical disease that in the opinion of the investigator could cause unacceptable safety risks or compromise compliance with the protocol e.g. impairment of gastrointestinal (GI) function, or GI disease that may significantly alter the absorption of the study drugs, uncontrolled diabetes
* Use of therapeutic coumarin derivatives (i.e. warfarin, acenoucumarol, phenprocoumon)
* Use of any medications that prolong the QT interval and CYP3A4 inhibitors if the treatment cannot be either safely discontinued or switched to a different medication prior to starting study drug administration. Please see www.qtdrugs.org for a comprehensive list of agents that prolong the QT interval as well as [Post-Text Supplement 2].
* Patients who have undergone major surgery ≤ 2 weeks prior to Visit 1 or who have not recovered from side effects of such surgery
* Patients who have received wide field radiotherapy ≤ 4 weeks or limited field radiation for palliation < 2 weeks prior to Visit 1 or who have not recovered from side effects of such therapy
* A history of noncompliance to medical regimens or inability or unwillingness to return for scheduled visits
* Patients who are pregnant, breast feeding or women of childbearing potential (WOCBP). Post-menopausal women must be amenorrheic for at least 12 months to be considered of non-childbearing potential Women of reproductive potential, to include female partners of heterosexual or bisexual patients, must agree to use an effective method of contraception during the study and for up to three months following termination of the study.
* Patients unwilling or unable to comply with the protocol

Eligibility criteria for patients from studies CAMN107G2301 or CAMN107DDE05 Patients currently participating in the Novartis-sponsored studies CAMN107G2301 or CAMN107DDE05 and benefiting from the nilotinib treatment according to the investigator will be offered the possibility to continue treatment with nilotinib in study CAMN107DDE06.

They will be included in study CAMN107DDE06 if the following criteria are fulfilled:

* Patient has an histologically confirmed diagnosis of GIST that is unresectable and/or metastatic
* Patient is currently enrolled in the studies CAMN107G2301 or CAMN107DDE05 in Germany and is on treatment with nilotinib
* Patient is currently benefiting from the treatment with nilotinib, as determined by the investigator
* Patient has demonstrated compliance, as assessed by the investigator, within the CAMN107G2301 or CAMN107DDE05 protocols requirements
* Patient has willingness and ability to comply with scheduled visits, treatment plans and any other study procedures
* Written informed consent obtained prior to enrollment in the study
* Pregnant or nursing (lactating) women, where pregnancy is defined as the state of a female after conception and until the termination of gestation, confirmed by a positive hCG laboratory test.
* Women of child-bearing potential, defined as all women physiologically capable of becoming pregnant, unless they are using highly effective methods of contraception during dosing and for 30 days of study medication. Highly effective contraception methods include:
* Total abstinence (when this is in line with the preferred and usual lifestyle of the subject. Periodic abstinence (e.g., calendar, ovulation, symptothermal, post-ovulation methods) and withdrawal are not acceptable methods of contraception

  * Female sterilization (have had surgical bilateral oophorectomy with or without hysterectomy) or tubal ligation at least six weeks before taking study treatment. In case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment
  * Male sterilization (at least 6 months prior to screening). For female subjects on the study the vasectomized male partner should be the sole partner for that subject.
  * Combination of any two of the following (a+b or a+c, or b+c):

    1. Use of oral, injected or implanted hormonal methods of contraception or other forms of hormonal contraception that have comparable efficacy (failure rate <1%), for example hormone vaginal ring or transdermal hormone contraception.
    2. Placement of an intrauterine device (IUD) or intrauterine system (IUS)
    3. Barrier methods of contraception: Condom or Occlusive cap (diaphragm or cervical/vault caps) with spermicidal foam/gel/film/cream/vaginal suppository

In case of use of oral contraception women should have been stable on the same pill for a minimum of 3 months before taking study treatment.

* Women are considered post-menopausal and not of child bearing potential if they have had 12 months of natural (spontaneous) amenorrhea with an appropriate clinical profile (e.g. age appropriate, history of vasomotor symptoms) or have had surgical bilateral oophorectomy (with or without hysterectomy) or tubal ligation at least six weeks ago. In the case of oophorectomy alone, only when the reproductive status of the woman has been confirmed by follow up hormone level assessment is she considered not of child bearing potential.
* Sexually active males unless they use a condom during intercourse while taking drug and for 30 days after stopping study medication and should not father a child in this period. A condom is required to be used also by vasectomized men in order to prevent delivery of the drug via seminal fluid.

Ages: 18 Years to 100 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 34 (Actual)
Dates: Start 2008-08-29 (Actual); Primary Completion 2024-12-18 (Actual); Study Completion 2024-12-18 (Actual)

CONTACTS AND LOCATIONS:
Overall Officials: Novartis Pharmaceuticals, Study Director — Novartis Pharmaceuticals
Locations (7):
- Novartis Investigative Site, Helsinki, Finland
- Novartis Investigative Site, Lyon, France
- Germany (4):
  - Novartis Investigative Site, Munich, Bavaria
  - Novartis Investigative Site, Bad Saarow
  - Novartis Investigative Site, Essen
  - Novartis Investigative Site, Hanover
- Novartis Investigative Site, Milan, MI, Italy

IPD SHARING:
Plan to Share IPD: Yes
Novartis is committed to sharing with qualified external researchers, access to patient-level data and supporting clinical documents from eligible studies. These requests are reviewed and approved by an independent review panel on the basis of scientific merit. All data provided is anonymized to respect the privacy of patients who have participated in the trial in line with applicable laws and regulations.
  This trial data availability is according to the criteria and process described on www.clinicalstudydatarequest.com
URL: https://www.clinicalstudydatarequest.com

RESULTS

PARTICIPANT FLOW:
Recruitment Details: Study consists of participants with unresectable or metastatic gastrointestinal stromal tumors (GIST) showing progression of disease from 5 countries: Germany, Spain, Finland, France, Italy
Pre-assignment Details: All enrolled participants received 400 mg bid dose of nilotinib.
Groups:
- Nilotinib: Participants who received 400 mg bid of nilotinib
Period: Core Phase
Arm/Group | Nilotinib
Started (All enrolled participants were included in the intent-to-treat (ITT) population and safety (SAF) population) | 41
Completed | 31
Not Completed | 10
Not completed — Adverse Event | 2
Not completed — Lack of Efficacy | 2
Not completed — Disease progression | 6
Period: Follow-Up Phase
Arm/Group | Nilotinib
Started | 31
Completed | 7
Not Completed | 24
Not completed — Missing values | 2
Not completed — Disease progression | 9
Not completed — Administrative problems | 3
Not completed — Lost to Follow-up | 1
Not completed — Withdrawal by Subject | 1
Not completed — Subject's condition no longer requires study drug | 1
Not completed — Adverse Event | 7

BASELINE CHARACTERISTICS:
Arm/Group | Nilotinib
Number analyzed (Participants) | 41
Age, Continuous [Mean (Standard Deviation); unit: Years] | 58 (10.4)
Sex: Female, Male [Count of Participants; unit: Participants]
  Female | 19
  Male | 22
Race/Ethnicity, Customized [Count of Participants; unit: Participants]
  Caucasian | 40
  Black | 1

OUTCOME MEASURES:

1. Primary Outcome: Proportion of Participants With Best Overall Response at Month 6 (Core Phase) Determined According to the RECIST v1.0.
Description: The primary efficacy measure is the proportion of patients reaching Complete Response (CR), Partial Response (PR), or Stable Disease (SD) by Month 6, as per RECIST v1.0. Definitions are as follows: CR requires at least two CRs at least four weeks apart before any progression; PR requires two or more PRs at least four weeks apart, without qualifying for CR; SD is at least one SD more than six weeks after treatment start, not qualifying for CR or PR. Progressive Disease (PD) is defined as progression or cancer-related death within 12 weeks of starting treatment, not qualifying for CR, PR, or SD. UNK refers to cases not meeting these criteria, such as absence of confirmed CR/PR, no SD after six weeks, or early progression. The percentage of patients with CR, PR, or SD will be presented with a one-sided exact 90% (or 80% two-sided) confidence interval for the ITT_F group.
Time Frame: from baseline to month 6, core phase
Population: The intent-to-treat (ITT) population consisted of all participants who received at least one dose of the study drug and had at least one post-baseline assessment of the primary efficacy variable (assessment according to RECIST). Participants without any post-baseline assessment of tumour were included if they were defined as progressive disease based on clinical evaluation.
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 41
Participants
  Complete Response (CR) | 0
  Partial Response (PR) | 14
  Stable Disease (SD) | 21
  Progressive Disease (PD) | 6
  Unknown (UNK) | 0

2. Secondary Outcome: Proportion of Participants With Objective Response Rate (ORR) at Month 6 (Core Phase) Observed According to RECIST
Description: Objective Response Rate (ORR) is defined as the proportion of patients in whom a complete (CR) or partial (PR) response was observed according to RECIST at month 6.
Time Frame: from baseline to month 6, core phase
Population: as for outcome 1
Measure: Number (80% Confidence Interval); unit: Percentage of responder
Arm/Group | Nilotinib
Number analyzed (Participants) | 41
Percentage of responder | 34.1 [24.2 to 45.3]

3. Secondary Outcome: Time to Response (TTR) at Month 6 (Core Phase)
Description: Time to response is defined as the time from start of treatment to the first objective tumor response (PR or CR) observed. Patients who did not achieve a confirmed PR or CR will be censored at last adequate tumor assessment date when they did not progress (including deaths not due to underlying disease).
Time Frame: from baseline to month 6, core phase
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nilotinib
Number analyzed (Participants) | 41
Days | 62 [57 to NA] — The upper bound of the confidence interval was not estimable due to insufficient events.

4. Secondary Outcome: Duration of Response (CR or PR) for Complete Study (Core and Follow-up Phases)
Description: Duration of response is defined as the time from onset of response (CR/PR) to objective tumor progression or death from any cause. Patients not experiencing progression or death will be censored with the date of their last adequate tumor assessment.
Time Frame: from date of first response (CR or PR) until progression or death, up to data cut off (up to approximately 16 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nilotinib
Number analyzed (Participants) | 21
Days | 2722 [588 to NA] — The upper bound of the confidence interval was not estimable due to insufficient events.

5. Secondary Outcome: Progression-free Survival (PFS) for Complete Study (Core and Follow-up Phases)
Description: Progression-free survival (PFS) is defined as the time from first study drug administration to objective tumor progression or death from any cause. If a patient has not had an event, PFS is censored at the date of last adequate tumor assessment. PFS will be explored graphically by presenting the Kaplan-Meier curve.
Time Frame: from date of first response (CR or PR) until progression or death, up to data cut off (up to approximately 16 years)
Population: as for outcome 1
Measure: Median (95% Confidence Interval); unit: Days
Arm/Group | Nilotinib
Number analyzed (Participants) | 31
Days | 2833 [791 to NA] — The upper bound of the confidence interval was not estimable due to insufficient events.

6. Secondary Outcome: Overall Survival for Complete Study (Core and Follow-up Phases)
Description: Overall Survival (OS) is defined as the time from first study drug administration to death from any cause. Participants alive at their last known follow-up were censored. No deaths occurred during the study.
Time Frame: from date of first response (CR or PR) until progression or death, up to data cut off (up to approximately 16 years)
Population: The intent-to-treat (ITT) population consisted of all participants who received at least one dose of the study drug.
Measure: Mean (Standard Deviation); unit: years
Arm/Group | Nilotinib
Number analyzed (Participants) | 41
years | NA (NA) — Overall survival could not be calculated due to an insufficient number of events

7. Secondary Outcome: Proportion of Participants With Treatment-emergent Adverse Events During the Entire Study (Core and Follow-up Phases)
Description: This measure summarizes the proportion of participants who experienced at least one treatment-emergent adverse event (TEAE) during the entire study period, including both core and follow-up phases. A TEAE was defined as an adverse event that began or worsened after the first dose of study treatment.
Time Frame: from the first dose through the end of the study (core and follow-up phases): including all visits up to the follow-up database lock (approximately 16 years)
Population: as for outcome 1
Measure: Count of Participants; unit: Participants
Arm/Group | Nilotinib
Number analyzed (Participants) | 41
Participants | 39

ADVERSE EVENTS:
Time Frame: Adverse events were collected from first dose through the end of the study (core and follow-up phases), including all visits up to the follow-up database lock (approximately 16 years).
Description: Any signs or symptoms were collected from first dose through the end of the study (core and follow-up phases), including all visits up to the follow-up database lock (approximately 16 years).
Groups:
- Total Core: Total Core phase
- Total Follow up: Total Follow up phase
Arm/Group | Total Core | Total Follow up
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/31
Serious Adverse Events (participants affected / at risk) | 10/41 | 14/31
Other Adverse Events (participants affected / at risk) | 39/41 | 28/31
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk:
Term (organ system) | Total Core (N=41) | Total Follow up (N=31)
MYOCARDIAL INFARCTION (Cardiac disorders) | 1 | 1
ABDOMINAL PAIN (Gastrointestinal disorders) | 2 | 2
DIARRHOEA (Gastrointestinal disorders) | 1 | 0
SUBILEUS (Gastrointestinal disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 0
PYREXIA (General disorders) | 2 | 2
HAEMOGLOBIN DECREASED (Investigations) | 1 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 0
TUMOUR RUPTURE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
ARTERIAL THROMBOSIS (Vascular disorders) | 1 | 0
CARDIAC FAILURE (Cardiac disorders) | 0 | 2
CARDIAC FAILURE CHRONIC (Cardiac disorders) | 0 | 1
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CARDIO-RESPIRATORY ARREST (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1
SUPRAVENTRICULAR TACHYCARDIA (Cardiac disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 2
VESTIBULAR DISORDER (Ear and labyrinth disorders) | 0 | 1
TOXIC NODULAR GOITRE (Endocrine disorders) | 0 | 1
GLAUCOMA (Eye disorders) | 0 | 1
OCULAR HYPERTENSION (Eye disorders) | 0 | 1
GENERAL PHYSICAL HEALTH DETERIORATION (General disorders) | 0 | 1
HYPERPLASIA (General disorders) | 0 | 1
VASCULAR STENT STENOSIS (General disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
MULTIPLE SCLEROSIS RELAPSE (Immune system disorders) | 0 | 1
INFECTION (Infections and infestations) | 0 | 1
SEPSIS (Infections and infestations) | 0 | 1
STREPTOCOCCAL SEPSIS (Infections and infestations) | 0 | 1
ARTERIAL RESTENOSIS (Injury, poisoning and procedural complications) | 0 | 1
KERATOACANTHOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PLASMA CELL MYELOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
HEADACHE (Nervous system disorders) | 0 | 1
NEURITIS (Nervous system disorders) | 0 | 1
DEPRESSION (Psychiatric disorders) | 0 | 1
ACUTE KIDNEY INJURY (Renal and urinary disorders) | 0 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PULMONARY HYPERTENSION (Respiratory, thoracic and mediastinal disorders) | 0 | 1
CIRCULATORY COLLAPSE (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
OTHER ADVERSE EVENTS (reported when occurring in more than 2% of participants in an arm); cells are participants affected of the arm's N at risk:
Term (organ system) | Total Core (N=41) | Total Follow up (N=31)
ANAEMIA (Blood and lymphatic system disorders) | 2 | 4
NEUTROPENIA (Blood and lymphatic system disorders) | 1 | 0
PALPITATIONS (Cardiac disorders) | 2 | 1
HYPOACUSIS (Ear and labyrinth disorders) | 1 | 1
GOITRE (Endocrine disorders) | 1 | 1
ABNORMAL SENSATION IN EYE (Eye disorders) | 1 | 0
DRY EYE (Eye disorders) | 1 | 1
EYELID PAIN (Eye disorders) | 1 | 1
OCULAR HYPERAEMIA (Eye disorders) | 1 | 0
ABDOMINAL PAIN (Gastrointestinal disorders) | 11 | 8
ABDOMINAL PAIN LOWER (Gastrointestinal disorders) | 1 | 1
ABDOMINAL PAIN UPPER (Gastrointestinal disorders) | 4 | 0
CONSTIPATION (Gastrointestinal disorders) | 7 | 9
DIARRHOEA (Gastrointestinal disorders) | 8 | 3
DYSPEPSIA (Gastrointestinal disorders) | 1 | 2
DYSPHAGIA (Gastrointestinal disorders) | 1 | 0
FLATULENCE (Gastrointestinal disorders) | 4 | 2
GASTRIC POLYPS (Gastrointestinal disorders) | 1 | 1
GASTRITIS EROSIVE (Gastrointestinal disorders) | 1 | 0
GASTROOESOPHAGEAL REFLUX DISEASE (Gastrointestinal disorders) | 2 | 1
HAEMORRHOIDS (Gastrointestinal disorders) | 1 | 1
HIATUS HERNIA (Gastrointestinal disorders) | 1 | 1
NAUSEA (Gastrointestinal disorders) | 8 | 5
TOOTHACHE (Gastrointestinal disorders) | 1 | 2
VOMITING (Gastrointestinal disorders) | 4 | 4
ASTHENIA (General disorders) | 11 | 2
CHEST DISCOMFORT (General disorders) | 1 | 0
CHEST PAIN (General disorders) | 1 | 0
FACE OEDEMA (General disorders) | 1 | 0
FATIGUE (General disorders) | 10 | 5
FEELING COLD (General disorders) | 2 | 1
LOCAL SWELLING (General disorders) | 1 | 0
MUCOSAL INFLAMMATION (General disorders) | 1 | 1
OEDEMA (General disorders) | 1 | 1
OEDEMA PERIPHERAL (General disorders) | 8 | 7
PYREXIA (General disorders) | 2 | 3
THIRST (General disorders) | 1 | 0
HEPATITIS TOXIC (Hepatobiliary disorders) | 1 | 0
HEPATOTOXICITY (Hepatobiliary disorders) | 3 | 1
HYPERBILIRUBINAEMIA (Hepatobiliary disorders) | 6 | 4
HYPERTRANSAMINASAEMIA (Hepatobiliary disorders) | 1 | 0
CYSTITIS (Infections and infestations) | 1 | 0
EAR INFECTION (Infections and infestations) | 1 | 0
FEBRILE INFECTION (Infections and infestations) | 1 | 0
GASTROENTERITIS (Infections and infestations) | 1 | 1
HERPES ZOSTER (Infections and infestations) | 1 | 1
NASOPHARYNGITIS (Infections and infestations) | 8 | 6
ORAL HERPES (Infections and infestations) | 1 | 0
RESPIRATORY TRACT INFECTION (Infections and infestations) | 1 | 0
TOOTH ABSCESS (Infections and infestations) | 1 | 1
TOOTH INFECTION (Infections and infestations) | 1 | 0
VIRAL INFECTION (Infections and infestations) | 1 | 1
ALANINE AMINOTRANSFERASE INCREASED (Investigations) | 2 | 3
BLOOD AMYLASE INCREASED (Investigations) | 1 | 0
BLOOD BILIRUBIN INCREASED (Investigations) | 1 | 2
BLOOD CREATININE INCREASED (Investigations) | 1 | 1
BLOOD GLUCOSE INCREASED (Investigations) | 1 | 1
GAMMA-GLUTAMYLTRANSFERASE INCREASED (Investigations) | 2 | 1
LIPASE INCREASED (Investigations) | 1 | 3
TRANSAMINASES INCREASED (Investigations) | 5 | 2
DECREASED APPETITE (Metabolism and nutrition disorders) | 5 | 0
HYPERCALCAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERCHOLESTEROLAEMIA (Metabolism and nutrition disorders) | 2 | 1
HYPERKALAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERLIPASAEMIA (Metabolism and nutrition disorders) | 1 | 1
HYPERURICAEMIA (Metabolism and nutrition disorders) | 1 | 0
HYPOPHOSPHATAEMIA (Metabolism and nutrition disorders) | 1 | 2
ARTHRALGIA (Musculoskeletal and connective tissue disorders) | 8 | 4
BACK PAIN (Musculoskeletal and connective tissue disorders) | 5 | 5
BONE PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
FLANK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 0
GROIN PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
JOINT SWELLING (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCLE SPASMS (Musculoskeletal and connective tissue disorders) | 5 | 5
MUSCLE TIGHTNESS (Musculoskeletal and connective tissue disorders) | 1 | 0
MUSCULOSKELETAL PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
MYALGIA (Musculoskeletal and connective tissue disorders) | 2 | 3
NECK PAIN (Musculoskeletal and connective tissue disorders) | 1 | 1
PAIN IN EXTREMITY (Musculoskeletal and connective tissue disorders) | 5 | 4
SKIN PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 2
SPINAL HAEMANGIOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 1 | 0
DIZZINESS (Nervous system disorders) | 2 | 3
DYSGEUSIA (Nervous system disorders) | 4 | 2
HEADACHE (Nervous system disorders) | 11 | 5
MEMORY IMPAIRMENT (Nervous system disorders) | 1 | 0
PARAESTHESIA (Nervous system disorders) | 1 | 5
PERIPHERAL SENSORY NEUROPATHY (Nervous system disorders) | 2 | 2
ANXIETY (Psychiatric disorders) | 2 | 1
ILLUSION (Psychiatric disorders) | 1 | 0
INSOMNIA (Psychiatric disorders) | 1 | 0
NERVOUSNESS (Psychiatric disorders) | 1 | 0
RESTLESSNESS (Psychiatric disorders) | 1 | 1
SLEEP DISORDER (Psychiatric disorders) | 1 | 1
HAEMATURIA (Renal and urinary disorders) | 2 | 0
NOCTURIA (Renal and urinary disorders) | 1 | 2
POLLAKIURIA (Renal and urinary disorders) | 2 | 1
RENAL FAILURE (Renal and urinary disorders) | 1 | 2
ERECTILE DYSFUNCTION (Reproductive system and breast disorders) | 2 | 1
NIPPLE OEDEMA (Reproductive system and breast disorders) | 1 | 0
NIPPLE PAIN (Reproductive system and breast disorders) | 1 | 0
PELVIC PAIN (Reproductive system and breast disorders) | 1 | 0
TESTIS DISCOMFORT (Reproductive system and breast disorders) | 1 | 0
COUGH (Respiratory, thoracic and mediastinal disorders) | 2 | 3
DYSPHONIA (Respiratory, thoracic and mediastinal disorders) | 1 | 1
DYSPNOEA (Respiratory, thoracic and mediastinal disorders) | 2 | 1
PLEURAL EFFUSION (Respiratory, thoracic and mediastinal disorders) | 1 | 3
THROAT IRRITATION (Respiratory, thoracic and mediastinal disorders) | 1 | 1
ALOPECIA (Skin and subcutaneous tissue disorders) | 8 | 9
DRY SKIN (Skin and subcutaneous tissue disorders) | 8 | 8
ECZEMA (Skin and subcutaneous tissue disorders) | 3 | 1
ERYTHEMA (Skin and subcutaneous tissue disorders) | 1 | 1
HYPERHIDROSIS (Skin and subcutaneous tissue disorders) | 2 | 1
NIGHT SWEATS (Skin and subcutaneous tissue disorders) | 1 | 1
PALMAR-PLANTAR ERYTHRODYSAESTHESIA SYNDROME (Skin and subcutaneous tissue disorders) | 2 | 2
PETECHIAE (Skin and subcutaneous tissue disorders) | 1 | 1
PHOTOSENSITIVITY REACTION (Skin and subcutaneous tissue disorders) | 1 | 2
PILOERECTION (Skin and subcutaneous tissue disorders) | 1 | 0
PRURITUS (Skin and subcutaneous tissue disorders) | 11 | 5
RASH (Skin and subcutaneous tissue disorders) | 10 | 6
XANTHELASMA (Skin and subcutaneous tissue disorders) | 1 | 1
ARTERIOSCLEROSIS (Vascular disorders) | 1 | 2
HOT FLUSH (Vascular disorders) | 2 | 1
HYPERTENSION (Vascular disorders) | 1 | 2
AGRANULOCYTOSIS (Blood and lymphatic system disorders) | 0 | 1
SPLENIC INFARCTION (Blood and lymphatic system disorders) | 0 | 1
ANGINA PECTORIS (Cardiac disorders) | 0 | 2
CARDIAC FAILURE CONGESTIVE (Cardiac disorders) | 0 | 1
CORONARY ARTERY DISEASE (Cardiac disorders) | 0 | 2
MITRAL VALVE INCOMPETENCE (Cardiac disorders) | 0 | 1
PERICARDIAL EFFUSION (Cardiac disorders) | 0 | 1
EAR SWELLING (Ear and labyrinth disorders) | 0 | 1
EXTERNAL EAR INFLAMMATION (Ear and labyrinth disorders) | 0 | 1
TINNITUS (Ear and labyrinth disorders) | 0 | 1
VERTIGO (Ear and labyrinth disorders) | 0 | 5
HYPERTHYROIDISM (Endocrine disorders) | 0 | 2
CONJUNCTIVAL HAEMORRHAGE (Eye disorders) | 0 | 1
EYE PAIN (Eye disorders) | 0 | 1
GLAUCOMA (Eye disorders) | 0 | 1
OCULAR HYPERTENSION (Eye disorders) | 0 | 1
PERIORBITAL OEDEMA (Eye disorders) | 0 | 1
ABDOMINAL DISCOMFORT (Gastrointestinal disorders) | 0 | 2
AEROPHAGIA (Gastrointestinal disorders) | 0 | 1
ASCITES (Gastrointestinal disorders) | 0 | 1
DIVERTICULUM INTESTINAL (Gastrointestinal disorders) | 0 | 1
DRY MOUTH (Gastrointestinal disorders) | 0 | 3
EPIGASTRIC DISCOMFORT (Gastrointestinal disorders) | 0 | 1
GASTRITIS HAEMORRHAGIC (Gastrointestinal disorders) | 0 | 1
GINGIVAL RECESSION (Gastrointestinal disorders) | 0 | 1
HAEMATOCHEZIA (Gastrointestinal disorders) | 0 | 1
LIP ULCERATION (Gastrointestinal disorders) | 0 | 1
REFLUX GASTRITIS (Gastrointestinal disorders) | 0 | 1
INFLAMMATION (General disorders) | 0 | 1
INFUSION SITE EXTRAVASATION (General disorders) | 0 | 1
MALAISE (General disorders) | 0 | 1
PSEUDOCYST (General disorders) | 0 | 1
CHOLELITHIASIS (Hepatobiliary disorders) | 0 | 1
HEPATIC PAIN (Hepatobiliary disorders) | 0 | 1
MULTIPLE SCLEROSIS (Immune system disorders) | 0 | 1
MULTIPLE SCLEROSIS RELAPSE (Immune system disorders) | 0 | 1
BRONCHITIS (Infections and infestations) | 0 | 2
CONJUNCTIVITIS (Infections and infestations) | 0 | 2
CORONAVIRUS INFECTION (Infections and infestations) | 0 | 1
EYE INFECTION (Infections and infestations) | 0 | 1
FOLLICULITIS (Infections and infestations) | 0 | 1
GANGRENE (Infections and infestations) | 0 | 1
GASTROINTESTINAL INFECTION (Infections and infestations) | 0 | 1
HERPES SIMPLEX (Infections and infestations) | 0 | 1
LOCALISED INFECTION (Infections and infestations) | 0 | 1
ONYCHOMYCOSIS (Infections and infestations) | 0 | 1
PERIODONTITIS (Infections and infestations) | 0 | 1
PNEUMONIA (Infections and infestations) | 0 | 1
RESPIRATORY TRACT INFECTION VIRAL (Infections and infestations) | 0 | 2
SINUSITIS (Infections and infestations) | 0 | 1
SKIN INFECTION (Infections and infestations) | 0 | 1
UPPER RESPIRATORY TRACT INFECTION (Infections and infestations) | 0 | 1
URINARY TRACT INFECTION (Infections and infestations) | 0 | 1
WOUND INFECTION (Infections and infestations) | 0 | 1
ARTHROPOD BITE (Injury, poisoning and procedural complications) | 0 | 1
CONTUSION (Injury, poisoning and procedural complications) | 0 | 1
FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
JOINT DISLOCATION (Injury, poisoning and procedural complications) | 0 | 1
RIB FRACTURE (Injury, poisoning and procedural complications) | 0 | 2
SKIN ABRASION (Injury, poisoning and procedural complications) | 0 | 1
SPLINTER (Injury, poisoning and procedural complications) | 0 | 1
THORACIC VERTEBRAL FRACTURE (Injury, poisoning and procedural complications) | 0 | 1
WOUND (Injury, poisoning and procedural complications) | 0 | 1
AMYLASE INCREASED (Investigations) | 0 | 3
ASPARTATE AMINOTRANSFERASE INCREASED (Investigations) | 0 | 1
C-REACTIVE PROTEIN INCREASED (Investigations) | 0 | 1
CARDIAC MURMUR (Investigations) | 0 | 1
COLONOSCOPY (Investigations) | 0 | 1
ELECTROCARDIOGRAM QT PROLONGED (Investigations) | 0 | 1
INTRAOCULAR PRESSURE INCREASED (Investigations) | 0 | 1
DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 1
FOLATE DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1
GOUT (Metabolism and nutrition disorders) | 0 | 1
HYPERAMYLASAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERGLYCAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERNATRAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPERPROTEINAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPOALBUMINAEMIA (Metabolism and nutrition disorders) | 0 | 1
HYPONATRAEMIA (Metabolism and nutrition disorders) | 0 | 2
IRON DEFICIENCY (Metabolism and nutrition disorders) | 0 | 2
TYPE 2 DIABETES MELLITUS (Metabolism and nutrition disorders) | 0 | 2
VITAMIN D DEFICIENCY (Metabolism and nutrition disorders) | 0 | 1
INTERVERTEBRAL DISC PROTRUSION (Musculoskeletal and connective tissue disorders) | 0 | 1
MUSCULAR WEAKNESS (Musculoskeletal and connective tissue disorders) | 0 | 2
MUSCULOSKELETAL CHEST PAIN (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOARTHRITIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOCHONDROSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
OSTEOLYSIS (Musculoskeletal and connective tissue disorders) | 0 | 1
BASAL CELL CARCINOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
HAEMANGIOMA OF BONE (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
PAPILLOMA (Neoplasms benign, malignant and unspecified (incl cysts and polyps)) | 0 | 1
CAROTID ARTERY STENOSIS (Nervous system disorders) | 0 | 1
CEREBROVASCULAR DISORDER (Nervous system disorders) | 0 | 1
DECREASED VIBRATORY SENSE (Nervous system disorders) | 0 | 1
DISTURBANCE IN ATTENTION (Nervous system disorders) | 0 | 1
HYPOAESTHESIA (Nervous system disorders) | 0 | 1
NYSTAGMUS (Nervous system disorders) | 0 | 1
PARESIS (Nervous system disorders) | 0 | 1
PARTIAL SEIZURES (Nervous system disorders) | 0 | 1
POLYNEUROPATHY (Nervous system disorders) | 0 | 2
VASCULAR DEMENTIA (Nervous system disorders) | 0 | 1
ANXIETY DISORDER (Psychiatric disorders) | 0 | 1
CONFUSIONAL STATE (Psychiatric disorders) | 0 | 1
MOOD SWINGS (Psychiatric disorders) | 0 | 1
PANIC ATTACK (Psychiatric disorders) | 0 | 1
BLADDER DISCOMFORT (Renal and urinary disorders) | 0 | 1
CALCULUS URINARY (Renal and urinary disorders) | 0 | 1
CHRONIC KIDNEY DISEASE (Renal and urinary disorders) | 0 | 2
DYSURIA (Renal and urinary disorders) | 0 | 1
URINARY RETENTION (Renal and urinary disorders) | 0 | 1
CATARRH (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EMPHYSEMA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
HIATUS HERNIA (Respiratory, thoracic and mediastinal disorders) | 0 | 1
PLEURITIC PAIN (Respiratory, thoracic and mediastinal disorders) | 0 | 1
SLEEP APNOEA SYNDROME (Respiratory, thoracic and mediastinal disorders) | 0 | 1
EYELID INFECTION (Skin and subcutaneous tissue disorders) | 0 | 1
HAIR COLOUR CHANGES (Skin and subcutaneous tissue disorders) | 0 | 1
NAIL DISORDER (Skin and subcutaneous tissue disorders) | 0 | 1
ONYCHOCLASIS (Skin and subcutaneous tissue disorders) | 0 | 1
SCAR PAIN (Skin and subcutaneous tissue disorders) | 0 | 1
STASIS DERMATITIS (Skin and subcutaneous tissue disorders) | 0 | 1
ASTRINGENT THERAPY (Surgical and medical procedures) | 0 | 1
GASTROOESOPHAGEAL REFLUX PROPHYLAXIS (Surgical and medical procedures) | 0 | 1
VITRECTOMY (Surgical and medical procedures) | 0 | 1
ANEURYSM (Vascular disorders) | 0 | 1
AORTIC ANEURYSM (Vascular disorders) | 0 | 1
HYPERTENSIVE CRISIS (Vascular disorders) | 0 | 1
INTERMITTENT CLAUDICATION (Vascular disorders) | 0 | 1
PERIPHERAL ARTERIAL OCCLUSIVE DISEASE (Vascular disorders) | 0 | 1
PERIPHERAL COLDNESS (Vascular disorders) | 0 | 1
VENOUS THROMBOSIS (Vascular disorders) | 0 | 1

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: Yes; Restriction type: Other
The terms and conditions of Novartis' agreements with its investigators may vary. However, Novartis does not prohibit any investigator from publishing. Any publications from a single-site are postponed until the publication of the pooled data (i.e., data from all sites) in the clinical trial.

DOCUMENTS (2):
  • Study Protocol (2018-11-26): https://cdn.clinicaltrials.gov/large-docs/09/NCT00756509/Prot_000.pdf
  • Statistical Analysis Plan (2025-03-17): https://cdn.clinicaltrials.gov/large-docs/09/NCT00756509/SAP_001.pdf